CLINICAL TRIAL: NCT07033403
Title: Effect of Low-Level Laser Therapy on Wound Healing and Post-extraction Pain Management of Primary Molars. (a Randomized Controlled Clinical Trial)
Brief Title: Effect of Low-Level Laser Therapy on Wound Healing and Post-extraction Pain Management of Primary Molars.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1002-11/2024
Record Dates: First submitted 2025-06-03; First posted 2025-06-24 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-06

CONDITIONS: Post-extraction Pain (PEP); Wound Healing
Keywords: wound healing; photobiomodulation; post-extraction pain (PEP)
MeSH Terms: interventions — Low-Level Light Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): intervention arm using low-level laser therapy photobiomodulation
  Interventions: Device: Low Level Laser Therapy
- placebo (Sham) (Placebo Comparator): sham (placebo) arm
  Interventions: Behavioral: Placebo plus Treatment As Usual

INTERVENTIONS:
Device: Low Level Laser Therapy — low-level laser therapy (LLLT) at a wavelength of 660nm (SiroLaser Blue, Dentsply Sirona, USA) after extraction
  Arms: intervention
Behavioral: Placebo plus Treatment As Usual — placebo (Sham) with only the aiming beam of thelow-level laser therapy (LLLT)
  Arms: placebo (Sham)

SUMMARY:
The goal of this clinical trial is to evaluate the effect of low-level laser therapy on wound healing of primary molar teeth extraction. in children aged 5-8 years with bilateral primary molars indicated for extraction. The main questions it aims to answer are:

* does low-level laser therapy affect wound healing of primary molar teeth extraction?
* does of low-level laser therapy affect post-extraction pain management of primary molar.? Researchers will compare placebo group (Sham side) to Intervention side ( split mouth design).

Participants will be subjected to low level laser and post-extraction instructions in the intervention side, while the placebo side will receive post-extraction instructions only, participants will come for follow up on days 3, and 7 after extraction, they will answer self-reported questionnare related to post-extraction pain , wound healing will also be measured from photographs of the extraction site using Image J soft-ware

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the effect of low-level laser therapy on wound healing of primary molar teeth extraction. in children aged 5-8 years with bilateral primary molars indicated for extraction. this is a split mouth randomized controlled clinical trial.

Each participant will have one side randomly assigned to intervention using low level diode laser at a wavelength of 660nm aimed at the extraction site 1 cm away for 60 seconds in continuous emission mode. the other side will be placebo side with just the aiming beam, in both visits the participant will be given post-extraction instructions

participants will come for follow up on days 3, and 7 after extraction, they will answer an arabic self-reported questionnaire comprising 33 items that assessed pain, discomfort, analgesic consumption, daily activities, and jaw-function impairment on the night of the extraction and after 7 days, wound healing will also be measured days 3 and 7 using of the extraction site using Wound healing index by Landry, Turnbull and Howley, and wound size will be measured using Image J soft-ware from the from photographs.

ELIGIBILITY:
Inclusion Criteria:

* • Age range from 5 - 8 years.

  * Children free of any systemic disease or special health care need.
  * No previous extractions.
  * Positive or definitely positive behaviour during preoperative assessments according to the Frankl Rating Scale (score 3 or 4).
  * Patients with bilateral primary molars indicated for extraction.
  * Patients whose parents will give their written consent to participate

Exclusion Criteria:

* Resorption more than one third of the root length.
* Signs of mobility.
* History of allergy to local anesthesia.
* Medical History involving conditions such as prolonged bleeding, platelet disorders, hypersensitivity, allergic reactions to pain relievers and contradictions to laser therapy.
* Acute pain.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
wound healing | days 3 and 7
  wound healing will be measured using using the Landry, Turnbull and Howley wound healing index , with minimum score 1 and maximum score 5 , as the score inceases this means better healing.
post-extraction pain (PEP) | days 3 and 7
  post- extraction pain will be measured using the Arabic Version of a self-reported Questionnaire Assessing Pain, Discomfort and Related Jaw Function Impairment in Children on the night of extraction and on day 7 using WONG-BAKER FACES pain scale with 0 minimum and 10 maximum value. the higher the value the worse the outcome.
wound size measurements | days 3 and 7
  wound size measurments immediately after the extraction, and at days 3 and using Image J software

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry-Alexandria University, Alexandria, Egypt